CLINICAL TRIAL: NCT01957956
Title: Pilot Clinical Trial of Allogeneic Tumor Lysate-Pulsed Autologous Dendritic Cell Vaccination in Newly Diagnosed Glioblastoma
Brief Title: Vaccine Therapy and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1272; NCI-2013-01743 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vaccine therapy and temozolomide) (Experimental): COURSE 1: Patients receive temozolomide PO daily on days 1-5.
  COURSES 2-3: Patients receive temozolomide PO daily on days 1-5 and malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on days 1, 3, and 5.
  COURSES 4-6: Patients receive temozolomide PO daily on days 1-5 and malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on day 1.
  COURSES 7-12: Patients receive malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on day 1.
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Malignant Glioma Tumor Lysate-Pulsed Autologous Dendritic Cell Vaccine; Drug: Temozolomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Malignant Glioma Tumor Lysate-Pulsed Autologous Dendritic Cell Vaccine — Given ID
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This pilot clinical trial studies vaccine therapy and temozolomide in treating patients with newly diagnosed glioblastoma. Vaccines made from a person's white blood cells mixed with tumor proteins may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vaccine therapy and temozolomide may be an effective treatment for glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of adjuvant temozolomide plus combined allogeneic tumor primary tumor culture lysate / autologous dendritic cell (DC) vaccination (malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine) in newly diagnosed glioblastoma patients following surgical debulking and external beam radiation therapy with concurrent temozolomide.

SECONDARY OBJECTIVES:

I. To document survival and progression-free survival in newly diagnosed glioblastoma patients receiving adjuvant temozolomide plus allogeneic tumor primary tumor culture lysate / autologous DC vaccination to historical data.

TERTIARY OBJECTIVES:

I. Determine the ability of allogeneic tumor primary tumor culture lysate / autologous DC vaccine to generate multiple tumor-associated antigens (TAA)-specific immune responses in newly diagnosed glioblastoma multiforme (GBM) patients.

II. Assess the relationship between ability tumor induce TAA-specific immune responses and evidence of immunosuppression (peripheral blood immunophenotyping by flow cytometry) following allogeneic tumor primary tumor culture lysate / autologous DC vaccine in newly diagnosed GBM patients.

III. Assess the relationship between efficacy endpoints (survival, progression-free survival, tumor response) and tumor-associated antigen immune response following combined autologous or allogeneic tumor lysate / DC vaccination and adjuvant temozolomide.

IV. Assess the relationship between efficacy endpoints (survival, progression-free survival, tumor response) and evidence of immunosuppression at baseline and over time with combined autologous or allogeneic tumor lysate / DC vaccination and adjuvant temozolomide.

OUTLINE:

COURSE 1: Patients receive temozolomide orally (PO) daily on days 1-5.

COURSES 2-3: Patients receive temozolomide PO daily on days 1-5 and malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine intradermally (ID) on days 1, 3, and 5.

COURSES 4-6: Patients receive temozolomide PO daily on days 1-5 and malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on day 1.

COURSES 7-12: Patients receive malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on day 1.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of undergoing apheresis for collection of mononuclear cells
* Histologically confirmed GBM (grade 4 astrocytoma) NOTE: gliosarcomas and other grade 4 astrocytoma variants (e.g., giant cell) may be included, primitive neuroectodermal tumor (PNET) variants are excluded; grade 4 oligodendrogliomas or oligoastrocytomas are specifically excluded
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500 / uL
* Platelets (PLT) >= 100,000 / uL
* Hemoglobin (HgB) >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper normal limit (UNL)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x UNL
* Creatinine =< 1 x UNL
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to understand and willingness to sign a written informed consent
* Willing to return to Mayo Clinic Rochester for follow-up
* Willing to provide tissue and blood samples for mandatory correlative research purposes
* Fixed or decreasing dose of corticosteroids (or no corticosteroids) >= 7 days prior to registration
* Completed standard external beam radiation with temozolomide
* Achieved a gross total or sub-total resection at time of surgery

Exclusion Criteria:

* Current or prior treatment for this cancer with immunotherapy and/or any other investigational agents
* Any of the following

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV), human T-cell lymphotropic virus (HTLV), hepatitis B (HepB), or hepatitis C (HepC) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of other malignancy including treated lower grade gliomas; EXCEPTIONS: non-melanotic skin cancer, carcinoma-in-situ of the cervix, or lower grade glioma that has never been treated previously; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 180 days (6 months), or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Active infection =< 5 days prior to registration or fever > 38 degrees Celsius (C) on day of registration
* History of tuberculosis or positive purified protein derivative (PPD) test
* Inability or unwillingness to have magnetic resonance imaging (MRI) scans performed (e.g. cardiac pacemaker-dependent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of significant toxicity, defined as grade 3 or higher adverse event that is possibly, probably, or definitely related to treatment measured using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 84 days
  Incidence of significant toxicity will be estimated by the number of patients with significant toxicity divided by the total number of evaluable patients.

SECONDARY OUTCOMES:
Change in immunologic correlates | Baseline to up to 5 years
  Change in immunologic correlates before and after vaccination treatment will be evaluated and summarized both quantitatively and graphically. Spearman rank correlation coefficient will be used to assess the correlations between baseline levels as well as between changes before and after treatment in these immunologic markers.
Clinical benefit rate | Up to 5 years
  The clinical benefit rate will be estimated by the number of patients with an objective status of stable disease (SD) for at least 12 months or an objective status of CR or PR at any time divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true clinical benefit rate will be calculated.
Duration of response | Up to 5 years
  Duration of response will be summarized descriptively.
Overall response rate | Up to 5 years
  The overall response rate will be estimated by the number of patients with an objective status of complete response (CR) or partial response (PR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Time to response | Up to 5 years
  Time to response will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Parney, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States